CLINICAL TRIAL: NCT02697656
Title: A Randomized Controlled Trial Assessing the Effectiveness of the Individual Placement and Support Model for Patients With Chronic Pain in an Outpatient Hospital Pain Clinic
Brief Title: The Effectiveness of Individual Placement and Support in Chronic Pain Patients
Acronym: IPSinPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Directorate of Health (Other Government); Norwegian Labour and Welfare Administration (Other)
Responsible Party: Principal Investigator, Silje Endresen Reme, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/14224
Record Dates: First submitted 2016-01-18; First posted 2016-03-03 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual + self-help (Active Comparator): Interdisciplinary treatment as usual at the outpatient pain clinic + an additional self-help binder with resources about pain management and employment advice.
  Interventions: Behavioral: Self-help; Behavioral: Treatment as usual
- Treatment as usual + IPS (Experimental): Individual job support (IPS) as an integrated part of the interdisciplinary treatment at the outpatient pain clinic.
  Interventions: Behavioral: IPS; Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: IPS — Individualized job support provided by an employment specialist
  Arms: Treatment as usual + IPS
Behavioral: Self-help — Self-help resources on obtaining employment and coping with chronic pain
  Arms: Treatment as usual + self-help
Behavioral: Treatment as usual — Transdisciplinary treatment at the pain clinic. This includes medical, psychological and physiotherapy treatment.

SUMMARY:
Individual Placement and support (IPS) is an evidence-based approach originally developed to help people with severe mental disorders to obtain and maintain employment. The effectiveness of IPS for patients with severe mental illness is well documented, but has never previously been tested for patients with chronic pain. In fact, employment support is rarely provided in pain clinics, despite an increasing focus on integrating work and health in all patient treatment (OECD, 2013). The aim of this study is to investigate the effectiveness of IPS as an integrated part of the interdisciplinary treatment for patients with chronic pain in a hospital outpatient clinic.

DETAILED DESCRIPTION:
Individual Placement and support (IPS) is an evidence-based approach originally developed to help people with severe mental disorders to obtain and maintain employment. IPS represents a relatively new approach to vocational rehabilitation and incorporates following principles: (1) Every person that wants to work, can work given that the person is provided with the appropriate work and environment. (2)The goal is employment in regular, competitive employment. (3) IPS is integrated with treatment. (4) Job search is individualised; based on the participants' preferences and competence. (5) Work incentives planning is provided; which includes counselling about how work can influence social security and other public benefits. The intention of this benefits counselling is to enable the participant to make informed decisions about work (job starts and changes). (6) The job support is not time-limited. (7) Finally, IPS differs from more traditional employment services in that it does not involve pre-vocational training, often referred to as "train, then place". (8) In IPS job search starts as soon as the client expresses an interest in work. Therefore, IPS follows the principle "place, then train".

The effectiveness of IPS for patients with severe mental illness is well documented. International research shows that IPS is more effective than other types of employment programs for this group of clients. However, the effect of IPS on patients with chronic pain in an outpatient hospital clinic is largely unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the pain clinic and eligible for interdisciplinary treatment
* Not currently working (long-term sick leave, disability pension or unemployed)
* Expressed desire to work

Exclusion Criteria:

* Living too far away from the pain clinic (outside of Oslo)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Competitive employment | At 12-months follow-up
  Hours/days/weeks worked in competitive employment the last 12 months

SECONDARY OUTCOMES:
Health-related quality of life | 6 and 12 months follow-up
  EQ5D termometer
Pain-related disability | 6 and 12 months follow-up
  Oswestry, modified to chronic pain patients
Pain intensity | 6 and 12 months follow-up
  Numeric Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Silje E Reme, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Silje Endresen Reme, Oslo, Norway

REFERENCES:
- [Background] Bond GR, Drake RE. Making the case for IPS supported employment. Adm Policy Ment Health. 2014 Jan;41(1):69-73. doi: 10.1007/s10488-012-0444-6. PMID 23161326
- [Background] Bond GR, Drake RE, Becker DR. An update on randomized controlled trials of evidence-based supported employment. Psychiatr Rehabil J. 2008 Spring;31(4):280-90. doi: 10.2975/31.4.2008.280.290. PMID 18407876
- [Derived] Sveinsdottir V, Jacobsen HB, Ljosaa TM, Linnemorken LTB, Knutzen T, Ghiasvand R, Reme SE. The Individual Placement and Support (IPS) in Pain Trial: A Randomized Controlled Trial of IPS for Patients with Chronic Pain Conditions. Pain Med. 2022 Sep 30;23(10):1757-1766. doi: 10.1093/pm/pnac032. PMID 35234931
- [Derived] Linnemorken LTB, Sveinsdottir V, Knutzen T, Rodevand L, Hernaes KH, Reme SE. Protocol for the Individual Placement and Support (IPS) in Pain Trial: A randomized controlled trial investigating the effectiveness of IPS for patients with chronic pain. BMC Musculoskelet Disord. 2018 Feb 13;19(1):47. doi: 10.1186/s12891-018-1962-5. PMID 29433493
- See also: The Study Protocol — http://www.ncbi.nlm.nih.gov/pubmed/29433493

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02697656/Prot_SAP_000.pdf